CLINICAL TRIAL: NCT01689987
Title: A Phase I Dose Escalation Study of Hydroxychloroquine With Infusional Cyclophosphamide, Pulse Dexamethasone and Rapamycin in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Hydroxychloroquine, Cyclophosphamide, Dexamethasone, and Sirolimus in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Emma Scott, Assistant Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00008296; NCI-2012-01754 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CR00022154; MR00041096; IRB00008296 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Hydroxychloroquine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (HCQ, sirolimus, cy/dex) (Experimental): Patients receive hydroxychloroquine PO daily on days 1-28 (days 5-28 of course 1), sirolimus PO on days -2 to 4, and cyclophosphamide IV continuously and dexamethasone PO on days 1-4. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Hydroxychloroquine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sirolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Hydroxychloroquine — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; RAPAMYCIN; SILA 9268A; WY-090217

SUMMARY:
This phase I trial studies the side effects and best dose of hydroxychloroquine when given together with cyclophosphamide, dexamethasone, and sirolimus in treating patients with multiple myeloma that has come back after a period of improvement or does not respond to treatment. Biological therapies, such as hydroxychloroquine, may stimulate the immune system in different ways and stop cancer cells from growing. Sirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, stopping them from dividing, or by stopping them from spreading. Giving hydroxychloroquine together with sirolimus, cyclophosphamide, and dexamethasone may be a better treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of hydroxychloroquine (HCQ) in combination with rapamycin (sirolimus) and infusional cyclophosphamide and pulse dexamethasone (cy/dex) for patients with relapsed/ refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate biological activity and efficacy of the combination of cyclophosphamide, dexamethasone, rapamycin and hydroxychloroquine in patients with relapsed/refractory multiple myeloma.

II. To determine whether this treatment regimen results in mammalian target of rapamycin (mTOR) and autophagy inhibition in primary myeloma cells during therapy and if this corresponds with treatment responses.

OUTLINE: This is a dose-escalation study of hydroxychloroquine.

Patients receive hydroxychloroquine orally (PO) daily on days 1-28 (days 5-28 of course 1), sirolimus PO on days -2 to 4, and cyclophosphamide intravenously (IV) continuously and dexamethasone PO on days 1-4. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed multiple myeloma
* Documented relapse or persistent disease after at least 1 prior therapy containing both bortezomib and lenalidomide; or at least 2 prior therapies containing bortezomib in one and lenalidomide in the other, or if intolerant of bortezomib and/or lenalidomide; prior autologous and allogeneic bone marrow transplantation are allowed
* Need for further treatment for myeloma, as determined by the patient's treating physician; this is defined as progression of clinical features (worsening anemia, renal function, bone disease, hypercalcemia, recurrent infections, and constitutional symptoms) OR biochemical progression (increasing M-spike in serum or urine, involved serum or urine free light chain over 2 consecutive time points greater than 4 weeks apart)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Ability to understand and the willingness to sign a written informed consent document
* Birth control is required with full barrier contraceptives or complete abstinence for the duration of time receiving therapy and for 6 months after completing the last drug taken
* The need for further treatment: this is defined as progression of clinical features (worsening anemia, renal function, bone disease, hypercalcemia, recurrent infections, and constitutional symptoms) OR biochemical progression (increasing M-spike in serum or urine, involved serum or urine free light chain over 2 consecutive time points greater than 4 weeks apart)

Exclusion Criteria:

* History of allergic reactions to compounds of similar chemical or biological composition to rapamycin or hydroxychloroquine
* Patients may not take any of the following medications while on study, but will be considered eligible if medication is discontinued at least 72 hours (hrs) prior to first dose of Rapamycin:

  * Carbamazepine
  * Rifabutin
  * Rifampin
  * Rifapentine
  * St. John's wort
  * Clarithromycin
  * Cyclosporine
  * Diltiazem
  * Erythromycin
  * Itraconazole
  * Fluconazole
  * Ketoconazole
  * Telithromycin
  * Verapamil
  * Voriconazole
  * Posaconazole
* Known macular degeneration or retinopathy (diabetic or otherwise), porphyria, or psoriasis (well-controlled psoriasis allowed provided under the care of a specialist who agrees to monitor the patient for exacerbations)
* Absolute neutrophil count (ANC) =< 1.0 x 10^9/L
* Platelets =< 50 x 10^9/L for any reason
* Serum creatinine >= 2.5 mg/dL
* Total or direct bilirubin >= 2.0 mg/dL
* Transaminases 2 x the upper limit of normal
* Fasting glucose >= 200 mg/dL
* Serum potassium < 3.4 mmol/l
* Serum phosphorus < 2.4 mg/dl
* Other conditions that would require therapy with hydroxychloroquine, including but not limited to, any of the following:

  * Systemic lupus
  * Rheumatoid arthritis
  * Porphyria cutanea tarda
  * Malaria treatment or prophylaxis
* Evidence of other active malignancy, except:

  * Basal cell or squamous cell carcinoma of the skin
  * Treated carcinoma in situ
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Uncontrolled ongoing infection
  * Human immunodeficiency virus (HIV)
  * Hepatitis B infection
  * Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
  * Active graft-versus-host disease (GvHD)
* Inability to understand or unwillingness to sign the informed consent document
* Concurrent anti-myeloma therapy within:

  * 7 days of prior corticosteroids
  * 14 days of prior antimyeloma agents, including thalidomide or lenalidomide
  * 28 days of a different investigational regimen
  * 14 days of any radiation
* Women of child-bearing who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 30 days after the last dose of study drug
* Women who are pregnant or breastfeeding
* History of G6PD deficiency
* Known history of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
MTD of hydroxychloroquine defined as the highest dose at which 0/6 or 1/6 subjects experience a dose limiting toxicity (DLT) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 | 56 days
  Incidence of DLTs will be tabulated for each dose level. Summarized using descriptive statistics or frequency distributions, as appropriate.

SECONDARY OUTCOMES:
Duration of overall response | Time that measurement criteria are met for response (whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented, assessed up to 12 months
  Will be summarized by 25th, 50th (median), and 75th percentile along with 95% confidence intervals using Kaplan-Meier method.
Myeloma response (stringent complete response, complete response, very good partial response, partial response, stable disease, and progressive disease), as assessed by the International Myeloma Working Group | Up to 12 months
  Presented with two-sided 95% exact binomial confidence interval.
Progression-free survival | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 12 months
  Will be summarized by 25th, 50th (median), and 75th percentile along with 95% confidence intervals using Kaplan-Meier method.
Time to response | Time from the first day of therapy until the time that measurement criteria are met for response, assessed up to 12 months
  Will be summarized by 25th, 50th (median), and 75th percentile along with 95% confidence intervals using Kaplan-Meier method.

OTHER OUTCOMES:
Mean percentage of p70S6 myeloma cells | Up to day 5 of course 2
  The mean percentage of p70S6 myeloma cells and the number of autophagic vesicles per bone marrow plasma cells will be compared between responders and non-responders using two-sample test if the data follows normal distribution or if the data does not follow normal distribution, transformation or non-parametric method will be considered.
Number of autophagic vesicles per bone marrow plasma cells | Up to day 5 of course 2
  The mean percentage of p70S6 myeloma cells and the number of autophagic vesicles per bone marrow plasma cells will be compared between responders and non-responders using two-sample test if the data follows normal distribution or if the data does not follow normal distribution, transformation or non-parametric method will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Scott, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States